CLINICAL TRIAL: NCT01636219
Title: Cough Efficiency in Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Daphna Vilozni, PhD, Head of Pediatric Pulmonary Laboratory, Sheba Medical Center
Other Study IDs: SHEBA-11-8709-OE-SMC
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Cystic Fibrosis
Keywords: Spirometry,; Cough
MeSH Terms: conditions — Cystic Fibrosis; Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The major causes of morbidity and mortality in Cystic Fibrosis (CF) are linked to the process of chronic inflammatory of the airway, leading to the progressive damage of the small bronchioles and subsequently to the proximal bronchi. A connection between weaknesses of respiratory muscles in CF and deficits of CFTR in the muscle has been established. Insufficient cough in CF patients may advance re-current respiratory infections. A voluntary cough flow volume (C-FVC) profile incorporates the characteristics of the forced expiratory flow volume curve (FE-VC). The study aims to explore the correspondence of voluntary cough-flow-volume and maximum expiratory flow-volume maneuvers in relation to disease complications in CF patients.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is the most common lethal life shortening genetic disease caused by mutations of the trans-membrane conductance regulator (CFTR) gene. The major causes of morbidity and mortality in CF are linked to the process of chronic inflammatory of the airway, leading to the progressive damage of the small bronchioles and subsequently to the proximal bronchi. Cough is a back-up mechanism for mucus clearance which comes into effect in health during emergency situations, such as following the inhalation of a foreign body, and in lung disease where often the primary host defense clearance mechanism, namely mucociliany clearance, is compromised

Several studies have showed a connection between weaknesses of respiratory muscles in CF and deficits of CFTR in the muscle; sustain infection of pseudomonas; lower than normal tension time index and low fat free mass [3-6]. Weakness of the respiratory muscle may insinuate insufficient cough in CF patients.

Effective cough is initiated in several mechanical stages: a) inhaling a variable amount of air, b) closure of the glottis, c) contraction of respiratory muscles, and d) forced expiration to residual volume [7-13] A voluntary cough flow volume (C-FVC) profile therefore, incorporates the characteristics of the forced expiratory flow volume curve (FEVC) in that the first "spike" represents the peak cough flow, and the volume exhaled by the cough corresponds with the vital capacity. The descending portion of the C-FVC including secondary spikes decrease in a linear fashion as lung volume goes down from total lung capacity to residual volume.10 similar to the FEVC flow decay. Any disturbance in either of the cough stages may impair its efficiency.

The aim of this study is to explore the information that can be gained on cough ability in a group of CF patients, by the performance of voluntary cough-flow-volume maneuver and in relation to the characteristics of a maximum expiratory flow-volume curve.

Study plan How does this advance the field? In this study we wish to evaluate for the first time the cough ability derived from the voluntary cough flow volume curve for detection of insufficient cough in patients with CF. We hope to show that the cough flow volume curve corresponds with changes in cough ability in these patients in relation to lung function deterioration.

What are the clinical implications? An objective following-up of cough ability deterioration may allow the opportunity to introduce special respiratory therapy for strengthening cough and ease secretion flow in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Cooperation with spirometry

Exclusion Criteria:

* exacerbation, patients younger than 8 years.

Ages: 8 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Any CF patient visiting the pulmonary function laboratory, above 8 years old, who could cooperate with spirometry and who had no exacerbation, upon signing agreement consent
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Cough flow volume indices compaired to healthy known data | 2 years
  The indices includs peak cough flow, Inspiratory capacity, number of cough spikes and cough vital capacity.

SECONDARY OUTCOMES:
forced vital capacity menuver | 2 years
  the cough flow volume curve is comapred to the forced vital capacity maneuver.

REFERENCES:
- [Background] Divangahi M, Matecki S, Dudley RW, Tuck SA, Bao W, Radzioch D, Comtois AS, Petrof BJ. Preferential diaphragmatic weakness during sustained Pseudomonas aeruginosa lung infection. Am J Respir Crit Care Med. 2004 Mar 15;169(6):679-86. doi: 10.1164/rccm.200307-949OC. Epub 2003 Dec 11. PMID 14670804
- [Background] Enright S, Chatham K, Ionescu AA, Unnithan VB, Shale DJ. The influence of body composition on respiratory muscle, lung function and diaphragm thickness in adults with cystic fibrosis. J Cyst Fibros. 2007 Nov 30;6(6):384-90. doi: 10.1016/j.jcf.2007.02.006. Epub 2007 Apr 2. PMID 17400035
- [Background] Divangahi M, Balghi H, Danialou G, Comtois AS, Demoule A, Ernest S, Haston C, Robert R, Hanrahan JW, Radzioch D, Petrof BJ. Lack of CFTR in skeletal muscle predisposes to muscle wasting and diaphragm muscle pump failure in cystic fibrosis mice. PLoS Genet. 2009 Jul;5(7):e1000586. doi: 10.1371/journal.pgen.1000586. Epub 2009 Jul 31. PMID 19649303
- [Background] Hayot M, Guillaumont S, Ramonatxo M, Voisin M, Prefaut C. Determinants of the tension-time index of inspiratory muscles in children with cystic fibrosis. Pediatr Pulmonol. 1997 May;23(5):336-43. doi: 10.1002/(sici)1099-0496(199705)23:53.0.co;2-i. PMID 9168507
- [Background] McCool FD, Leith DE. Pathophysiology of cough. Clin Chest Med. 1987 Jun;8(2):189-95. PMID 3621873
- [Background] Beardsmore CS, Wimpress SP, Thomson AH, Patel HR, Goodenough P, Simpson H. Maximum voluntary cough: an indication of airway function. Bull Eur Physiopathol Respir. 1987 Sep-Oct;23(5):465-72. PMID 3450329
- [Background] Pedersen OF, Lyager S, Ingram RH Jr. Airway dynamics in transition between peak and maximal expiratory flow. J Appl Physiol (1985). 1985 Dec;59(6):1733-46. doi: 10.1152/jappl.1985.59.6.1733. PMID 4077782
- [Background] Langlands J. The dynamics of cough in health and in chronic bronchitis. Thorax. 1967 Jan;22(1):88-96. doi: 10.1136/thx.22.1.88. No abstract available. PMID 6031920
- [Background] Bianchi C, Baiardi P. Cough peak flows: standard values for children and adolescents. Am J Phys Med Rehabil. 2008 Jun;87(6):461-7. doi: 10.1097/PHM.0b013e318174e4c7. PMID 18496248